CLINICAL TRIAL: NCT01110720
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety and Efficacy of Davunetide for the Treatment of Progressive Supranuclear Palsy
Brief Title: Study to Evaluate the Safety and Efficacy of Davunetide for the Treatment of Progressive Supranuclear Palsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-108-231
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — davunetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Davunetide 30 mg BID (Experimental)
  Interventions: Drug: Davunetide
- Placebo (Placebo Comparator)
  Interventions: Drug: Davunetide; Drug: Placebo

INTERVENTIONS:
Drug: Davunetide — Davunetide Nasal Spray 30 mg BID IN 52 weeks
Drug: Placebo — Placebo Nasal Spray BID IN 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of davunetide for the treatment of Progressive Supranuclear Palsy.

DETAILED DESCRIPTION:
A Phase 2/3,Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Davunetide for the Treatment of Progressive Supranuclear Palsy

ELIGIBILITY:
Inclusion Criteria:

* Probable or possible PSP defined as:

  * at least a 12-month history of postural instability or falls during the first 3 years that symptoms are present; and
  * at screening, a decreased downward saccade velocity defined as observable eye movement (deviation from the "main sequence" linear relationship between saccade amplitude and saccade velocity) or, supranuclear ophthalmoplegia defined as 50% reduction in upward gaze or 30% reduction in downward gaze; and
  * age at symptom onset of 40 to 85 years by history; and
  * an akinetic-rigid syndrome with prominent axial rigidity.
* Aged 41 to 85 years at the time of screening.
* Judged by investigator to be able to comply with neuropsychological evaluation at baseline and throughout the study.
* Must have reliable caregiver accompany subject to all study visits. Caregiver must read, understand, and speak local language fluently to ensure comprehension of informed consent form and informant-based assessments of subject. Caregiver must also have frequent contact with subject (at least 3 hours per week at one time or at different times) and be willing to monitor study medication compliance and the subject's health and concomitant medications throughout the study.
* Modified Hachinski score ≤ 3 (Appendix 7). This modified Hachinski will not include the focal neurological signs, symptoms or pseudobulbar affect questions, given the prominence of all 3 in PSP.
* Score ≥ 15 on the mini-mental state examination (MMSE) at screening (Visit 1).
* Written informed consent provided by subject (or legally-appointed representative, as appropriate) and caregiver (if not the legally-appointed representative) who are both fluent local language speakers.
* Subject resides outside a skilled nursing facility or dementia care facility at the time of screening, and admission to such a facility is not planned. Residence in an assisted living facility is allowed.
* If the subject is receiving levodopa/carbidopa, levodopa/benserazide, a dopamine agonist, catechol-o-methyltransferase (COMT) inhibitor, or other Parkinson's medication,with teh exception of Azilect(rasagiline), the dose must have been stable for at least 60 days prior to the screening visit (Visit 1) and must remain stable for the duration of the study. No such medication can be initiated during the study. Subjects receiving rasagiline or CoQ10 must be on a stable dose for at least 90 days prior to the screening visit.
* Able to tolerate the MRI scan during screening with either no sedation or low dose lorazepam.
* Able to ambulate independently or with assistance defined as the ability to take at least 5 steps with a walker (guarding is allowed provided there is no contact) or the ability to take at least 5 steps with the assistance of another person who can only have contact with one upper extremity.
* Presence of symptoms for less than 5 years or the presence of symptoms for more than 5 years with a PSPRS baseline score ≥ 40.
* Stable on all other chronic medications for at least 30 days prior to the screening visit (Visit 1).

Exclusion Criteria:

* Insufficient fluency in local language to complete neuropsychological and functional assessments.
* A diagnosis of Amyotrophic Lateral Sclerosis or other motor neuron disease.
* Any of the following:

  * Abrupt onset of symptoms defined in inclusion criteria 1 associated with ictal events,
  * Head trauma related to onset of symptoms defined in inclusion criteria 1,
  * Severe amnesia within 6 months of the symptoms defined in inclusion criteria 1,
  * Cerebellar ataxia,
  * Choreoathetosis,
  * Early, symptomatic autonomic dysfunction; or
  * Tremor while at rest.
* Presence of other significant neurological or psychiatric disorders including (but not limited to) Alzheimer's disease; dementia with Lewy bodies; prion disease; Parkinson's disease (which has not subsequently been revised to PSP); any psychotic disorder; severe bipolar or unipolar depression; seizure disorder; tumor or other space-occupying lesion; or history of stroke or head injury with loss of consciousness for at least 15 minutes within the past 20 years.
* Within 4 weeks of screening or during the course of the study, concurrent treatment with memantine; acetylcholinesterase inhibitors; antipsychotic agents (other than quetiapine) or mood stabilizers (e.g., valproate, lithium); or benzodiazepines (except as below).

  * Low dose lorazepam (not more than 2 mg) may be used for sedation prior to MRI scans for those subjects requiring sedation. Neuropsychological testing may not be performed after lorazepam administration.
  * Subjects who take short acting benzodiazepines (only temazepam or zolpidem are allowed) for sleep may continue to do so if they have been on a stable dose for 30 days prior to screening.
  * Clonazepam may be used for treatment of dystonia or painful rigidity associated with PSP if the dose has been stable for 90 days prior to screening and is not expected to change during the course of the study.
* Treatment with lithium, methylene blue, tramiprosate, ketone bodies, latrepirdine, or any putative disease-modifying agent directed at tau within 90 days of screening.
* A history of alcohol or substance abuse within 1 year prior to screening and deemed to be clinically significant by the site investigator.
* Any malignancy (other than non-metastatic dermatological conditions) within 5 years of the screening visit (Visit 1) or current clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disease. For the non-cancer conditions, if the condition has been stable for at least one year before the screening visit and is judged by the site investigator not to interfere with the subject's participation in the study, the subject may be included.
* Clinically significant laboratory abnormalities at screening, including creatinine ≥ 2.5 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times the upper limit of the normal reference range, vitamin B12 below the laboratory normal reference range, or thyroid stimulating hormone TSH above laboratory normal reference range.
* The systolic blood pressure measurement is > 190 or < 85 mm Hg. The diastolic blood pressure measurement is > 105 or < 50 mm Hg at screening.
* Abnormal ECG tracing at screening and judged to be clinically significant by the site investigator.
* Treatment with any investigational drugs or device within 90 days of screening.
* Known history of serum or plasma progranulin level less than one standard deviation below the normal subject mean for the laboratory performing the assay.
* Known presence of known disease-associated mutation in TDP-43, PGRN, CHMPB2, or VCP genes or any other frontotemporal lobar degeneration (FTLD) causative genes not associated with underlying tau pathology (e.g., Chromosome 9 associated FTD).
* History of deep brain stimulator (DBS) surgery other than sham surgery for DBS clinical trial.
* History of early, prominent rapid eye movement (REM) sleep behavior disorder.
* Women who are pregnant or lactating and women of childbearing potential who are not using at least two different forms of medically recognized and highly effective methods of birth control, resulting in a low failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* An employee or relative of an employee of the Sponsor, a clinical site, or Contract Research Organization participating in the study.
* Significant anatomical nasal abnormality (e.g., septal deviation obstructing airflow to at least one nostril or septal perforation) or history of nasal turbinate surgery.
* History of a clinically significant medical condition that would interfere with the subject's ability to comply with study instructions, would place the subject at increased risk, or might confound the interpretation of the study results.
* Contraindication to MRI examination for any reason (e.g., severe claustrophobia, ferromagnetic metal in body).
* Structural abnormality on MRI that precludes diagnosis of PSP, such as cortical infarct in brain region that might account for subject's symptoms.
* In subjects receiving anti-Parkinson's Disease medication at the time of screening, in the opinion of the investigator substantial worsening of motor signs or symptoms compared with normal functioning following overnight withdrawal of the anti-Parkinson medication.
* Known hypersensitivity to davunetide or any ingredient of the formulation.

Ages: 41 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Efficacy, as measured by change from baseline scores of the Progressive Supranuclear Palsy Rating Scale (PSPRS) at 52 weeks | 52 weeks
Efficacy, as measured by the change from baseline of the Schwab and England Activities of Daily Living Scale (SEADL) at 52 weeks | 52 weeks
Safety, as measured by reported AEs, electrocardiograms (ECG), nasal examinations and clinical laboratory measures | 52 weeks

SECONDARY OUTCOMES:
Efficacy, as measured by the Clinical Global Impression of Change (CGI-C) at 52 weeks | 52 weeks
Brain atrophy, as measured by change from baseline of ventricular volumes measured by volumetric brain MRI at 52 weeks. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, M.D., PhD., Principal Investigator — Memory and Aging Center, University of California, San Francisco
Locations (48):
- United States (28):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Muhammed Ali Parkinson Center and Movement Disorders Clinic, Phoenix, Arizona
  - Mayo Clinic, AZ, Scottsdale, Arizona
  - USC Keck School of Medicine, Los Angeles, California
  - David Geffen School of Medicine - UCLA, Los Angeles, California
  - UCSD/VA Neurology Service, San Diego, California
  - UCSF Memory and Aging Center, San Francisco, California
  - Colorado Neurological Institute - Rocky Mountain Movement Disorders Ctr, PC, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Mayo Clinic, Florida, Jacksonville, Florida
  - The Frances J. Zesiewicz Foundation for Parkinson's Disease at USF, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Medical Center Parkinson Disease & Movement Disorders Center, Kansas City, Kansas
  - University of Louisville Division of Movement Disorders, Louisville, Kentucky
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota Department of Neuology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, MN, Rochester, Minnesota
  - UMDNJ - Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - Univeristy of North Carolina Department of Neurology, Chapel Hill, North Carolina
  - University Hospitals Case Medical CenterNI Movement Disorders Center, South Euclid, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Center for Alzheimer's Care, Imaging &Research, Salt Lake City, Utah
- The Alfred Hospital, Melbourne, Victoria, Australia
- Canada (5):
  - London Sciences Health Center University Hospital, London, Ontario
  - Parkinson's Disease & Movement Disorders Clinic, Ottawa, Ontario
  - Toronto Western Hospital University Health Network, Toronto, Ontario
  - CHUM-Notre Dame Hospital Unité de Troubles du Mouvement, Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
- France (3):
  - Limoges University Hospital, Limoges
  - Hopital Timone, Marseille
  - Hôpitaux de Paris, Paris
- Germany (8):
  - Humboldt University Charité, Berlin
  - Neurologisch Klinik der Ruhr-Universität im St. Josef-Hospital, Bochum
  - Universitätsklinikum Carl Carus an der Technischen Universität, Dresden
  - Paracelsus-Elena Klinik, Kassel
  - Philipps Universität Marburg, Marburg
  - Klinikum Großhadern, München
  - Universität Rostock Zentrum für Nervenheilkunde und Poliklinik, Rostock
  - Universitäts- und Rehabilitationskliniken Ulm, Ulm
- United Kingdom (3):
  - Princess Royal Hospital, Haywards Heath
  - Clinical Ageing Research Unit (CARU) Newcastle University, Newcastle
  - Greater Manchester Neuroscience Centre, Salford

REFERENCES:
- [Derived] Hoglinger GU, Schope J, Stamelou M, Kassubek J, Del Ser T, Boxer AL, Wagenpfeil S, Huppertz HJ; AL-108-231 Investigators; Tauros MRI Investigators; Movement Disorder Society-Endorsed PSP Study Group. Longitudinal magnetic resonance imaging in progressive supranuclear palsy: A new combined score for clinical trials. Mov Disord. 2017 Jun;32(6):842-852. doi: 10.1002/mds.26973. Epub 2017 Apr 24. PMID 28436538
- [Derived] Boxer AL, Lang AE, Grossman M, Knopman DS, Miller BL, Schneider LS, Doody RS, Lees A, Golbe LI, Williams DR, Corvol JC, Ludolph A, Burn D, Lorenzl S, Litvan I, Roberson ED, Hoglinger GU, Koestler M, Jack CR Jr, Van Deerlin V, Randolph C, Lobach IV, Heuer HW, Gozes I, Parker L, Whitaker S, Hirman J, Stewart AJ, Gold M, Morimoto BH; AL-108-231 Investigators. Davunetide in patients with progressive supranuclear palsy: a randomised, double-blind, placebo-controlled phase 2/3 trial. Lancet Neurol. 2014 Jul;13(7):676-85. doi: 10.1016/S1474-4422(14)70088-2. Epub 2014 May 27. PMID 24873720